CLINICAL TRIAL: NCT02711241
Title: Optimal Analgesia in Acute Gastroenteritis in Emergency Department Setting: Dipyrone Versus Papaverine
Brief Title: Optimal Analgesia in Acute Gastroenteritis
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Not enough patients
Sponsor: Hadassah Medical Organization (Other)
Responsible Party: Principal Investigator, STALNIKOWICZ-DARVASI RUTH, Professsor, Hadassah Medical Organization
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AGE123-HMO-CTIL
Record Dates: First submitted 2011-03-01; First posted 2016-03-17 (Estimated); Last update posted 2016-03-17 (Estimated); Status verified 2016-03

CONDITIONS: Gastroenteritis
Keywords: Gastroenteritis; Analgesia; Emergency department
MeSH Terms: conditions — Gastroenteritis; Agnosia; Emergencies | interventions — Dipyrone; Papaverine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Dipyrone (Active Comparator)
  Interventions: Drug: Dipyrone
- Papaverine (Active Comparator)
  Interventions: Drug: Papaverine

INTERVENTIONS:
Drug: Dipyrone — 1 gram by slow IV infusion
  Other Names: Optalgin
  Arms: Dipyrone
Drug: Papaverine — 80 mg by slow intravenous infusion
  Arms: Papaverine

SUMMARY:
The purpose of this study is to find out an optimal way of analgesia in case of acute infectious gastroenteritis the investigators are going to compare two medicines that are used on everyday basis (without being ever before subject to scientifical study): Dipyrone and papaverine The study is done in the Emergency Department setting. Thus, only first 6 hours of treatment is included in study

ELIGIBILITY:
Inclusion Criteria:

* acute gastroenteritis
* VAS scale of pain perception at least 4

Exclusion Criteria:

* pregnancy
* allergy to any one of study preparations
* blood pressure less than 85 on admission
* surgical condition (acute abdomen) suspected or diagnosed

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2010-06; Primary Completion 2010-12 (Actual); Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
Change in pain assessment (VAS) as opposed the pain assessment on admission | 30 min, 1 hour, 2 hours, on discharge (up to 24 hours)

SECONDARY OUTCOMES:
Need for second analgesic medicine | 24 hours

CONTACTS AND LOCATIONS:
Overall Officials: Ruth Stanikowitz, MD, Principal Investigator — Hadassah Medical Organization
Locations (1):
- Hadssah Medical Organisation, Jerusalem, Israel